CLINICAL TRIAL: NCT01270594
Title: A Pilot Study to Evaluate a Telepharmacy Intervention to Improve Inhaler Adherence in Veterans With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: William S. Middleton Memorial Veterans Hospital (U.S. Federal Agency); American Society of Health-System Pharmacists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-2010-1187
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD Counseling Intervention (Experimental): Pharmacist counseling intervention delivered via telephone.
  Interventions: Behavioral: COPD Inhaler Counseling
- Usual Care (Other)
  Interventions: Behavioral: Usual Pharmacy Care

INTERVENTIONS:
Behavioral: COPD Inhaler Counseling — The counseling will be performed via telephone by a pharmacist at the William S Middleton Memorial Veterans Hospital. The counseling will include education about inhaled COPD medication, inhaler technique review, reminder tools, and motivational interviewing.
  Arms: COPD Counseling Intervention
Behavioral: Usual Pharmacy Care — The usual care arm will receive standard care from the William S Middleton Memorial Veterans Hospital pharmacists.
  Arms: Usual Care

SUMMARY:
Hypothesis: Can a counseling intervention, delivered by a pharmacist, increase inhaler adherence in veterans with COPD who have demonstrated poor inhaler adherence through pharmacy refill records?

Veterans who receive who receive daily maintenance inhalers from the William S Middleton Memorial Veterans Hospital Pharmacy and who have a medication possession ratio less than 80% over the previous six months will be invited to participate in the study. This study will randomize 100 participants to a usual care arm or a pharmacist counseling intervention. Final data collection will be six months after randomization to determine if both self-reported and refill record adherence has changed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans established with the William S. Middleton Memorial Veterans Hospital and associated Community Based Outpatient Clinics
* Fill their inhaled COPD medications with the VHA
* A diagnosis of COPD and an active prescription for a twice daily long-acting beta-agonist and/or long-acting anticholinergic with or without a prescription for inhaled corticosteroids for at least 4 months.
* Non-adherence to at least one COPD medication, a medication possession ratio of less than 80% or over 120% via the pharmacy refill records.

Exclusion Criteria:

* Patients with a diagnosis or electronic medical record note regarding significant hearing impairment.
* Patients with a diagnosis regarding cognitive deficit and activated power of attorney.
* Patients who use daily nebulization instead of inhalers for maintenance medication.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Adherence to daily inhaled COPD medications | Previous six months
  Adherence will be measured by pharmacy refill records and by participant self-report

SECONDARY OUTCOMES:
COPD exacerbations | Previous six months
  Participants will be asked how many episodes of worsening their COPD has required additional medical care and/or the use of an oral steroid or antibiotic.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Schuna, RPh MS, Principal Investigator — William S. Middleton Memorial Veterans Hospital
Locations (1):
- UW-Madison School of Pharmacy, Madison, Wisconsin, United States